CLINICAL TRIAL: NCT00420082
Title: A Randomized, Double-Blind, 4 Way Cross-over, Placebo Controlled Trial to Evaluate the Onset of Action of Bilastine 20 mg vs. Placebo, Cetirizine 10 mg, and Fexofenadine 120 mg in the Vienna Challenge Chamber
Brief Title: A Randomized, Double-Blind, 4-way Crossover Study to Evaluate the Efficacy of Bilastine in the Vienna Challenge Chamber
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BILA-2306/ACC; 2006-003004-19 (EudraCT Number)
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Rhinitis; Seasonal; Allergic; Pollen allergy; Environmental Exposure Chamber; Challenge Chamber
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis | interventions — bilastine; fexofenadine; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Bilastine 20 mg
  Interventions: Drug: Bilastine
- 2 (Active Comparator): Fexofenadine 120 mg
  Interventions: Drug: Fexofenadine
- 3 (Active Comparator): Cetirizine 10 mg
  Interventions: Drug: Cetirizine
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bilastine — Encapsulated Bilastine 20 mg tablets Q.D.
  Arms: 1
Drug: Fexofenadine — Encapsulated Fexofenadine 120 mg tablets Q.D.
  Other Names: Allegra
  Arms: 2
Drug: Cetirizine — Encapsulated Cetirizine 10 mg tablets Q.D.
  Other Names: Zyrtec
  Arms: 3
Drug: Placebo — Encapsulated Placebo tablets Q.D.
  Arms: 4

SUMMARY:
This is a randomized, double blind, active and placebo controlled, 4 way crossover study in patients with seasonal allergic rhinitis. Patients will receive a single dose of bilastine 20 mg, Cetirizine 10 mg, Fexofenadine 120 mg, and placebo in the Vienna Challenge Chamber.

DETAILED DESCRIPTION:
The objective of the study is to determine the effect of a single dose of bilastine 20 mg on nasal symptoms of allergic rhinitis provoked by spending 4 hours in the Vienna Challenge Chamber . This effect will be compared to that action of Cetirizine 10 mg, Fexofenadine 120 mg, and placebo. To explore the onset of action, patients will receive study drug two hours after the start of the provocation on Day 1.Patients will remain in theVCC for an additional four hours. On Day 2, patients will return to the VCC post-dose hours 22-26.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of seasonal allergic rhinitis
* Have a positive (as defined in the protocol) skin prick or RAST test within 12 months prior to the screening visit

Exclusion Criteria:

* Have a clinically significant illness or disease
* Have unstable asthma
* Has participated in a clinical trial 30 days prior to the screening visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2006-10; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Onset of action and action duration

SECONDARY OUTCOMES:
Nasal and ocular symptom scores
Nasal airflow resistance
Nasal secretion weight
FEV1
Routine safety parameters (vital signs, ECGs, clinical laboratory tests)

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Horak, Professor, Principal Investigator — ENT University Clinic Vienna
Locations (1):
- Allergy Center Vienna West, Vienna, Austria

REFERENCES:
- [Result] Horak F, Zieglmayer P, Zieglmayer R, Lemell P. The effects of bilastine compared with cetirizine, fexofenadine, and placebo on allergen-induced nasal and ocular symptoms in patients exposed to aeroallergen in the Vienna Challenge Chamber. Inflamm Res. 2010 May;59(5):391-8. doi: 10.1007/s00011-009-0117-4. Epub 2009 Nov 27. PMID 19943178